CLINICAL TRIAL: NCT01617473
Title: Randomized Trial of Unmanipulated Mobilized Blood/Marrow Versus Blood Haploidentical Transplant With Standard-risk Leukemia
Brief Title: Randomized Trial of Mobilized Blood/Marrow Versus Blood Transplant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: patients' reluctance
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang, chief of peking university institute of hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PUPH IRB [2012] (27)
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Transplantation

ARMS (2):
- procedure/surgery (Experimental): transplant with G-CSF mobilized PBSCs
  Interventions: Procedure: transplant with PBSCs
- other (No Intervention): no intervention after transplant with mobilized BMPB

INTERVENTIONS:
Procedure: transplant with PBSCs — mobilized PBSCs for 2 consecutive days
  Other Names: G-CSF mobilized peripheral blood stem cells
  Arms: procedure/surgery

SUMMARY:
The use of peripheral blood stem cells(PBSCs) is rapidly growing in the allogeneic transplantation setting as an alternative to bone marrow (BM).It was found that the use of PBSCs is associated with faster hematologic recovery but have yielded differing results regarding the incidence of graft-versus-host-disease (GVHD) and relapse.

The study hypothesis:

transplantation of mobilized PBSC to haploidentical donor with standard-risk leukemia had comparable engraftment and non-relapse mortality to mobilized BM combined with PBSCs

DETAILED DESCRIPTION:
The donors were primed with granulocyte-colony stimulating factor (G-CSF) injected subcutaneously for five consecutive days. In the trial group, the PBSCs were harvested on the fourth and fifth day;in the control group, the bone marrow cells were harvested on the fourth day and the PBSCs were harvested on the fifth day.

ELIGIBILITY:
Inclusion Criteria:

* Standard risk of Recipients of haploidentical stem cell transplantation with myeloablative conditioning regimens

Exclusion Criteria:

* Active, uncontrolled infection

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
incidence of engraftment | paticipants will be followed for the duration of hospital stay,an expected average of 30 days
  number of participants with engraftment at 30d

SECONDARY OUTCOMES:
incidence of non-relapse mortality | 1 year
  number of participants with non-relapse mortality at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, M.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People'S Hospital, Beijing, China